CLINICAL TRIAL: NCT06746649
Title: Healthy Aging: Effects of Time-specific Exercise on Functional, Structural, Metabolic and Immune Parameters in Circadian Context
Brief Title: Time-specific Exercise in Circadian Context
Acronym: CAEx
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Comenius University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APVV-21-0164
Record Dates: First submitted 2024-06-11; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Osteopenia; Osteoporosis; Aging
Keywords: bone mineral density; circadian rhythm; elderly
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis

STUDY DESIGN:
Intervention Model Description: In total, 34 previously untrained elderly subjects of both sexes, age range 65 - 80-year-old, will be recruited according to inclusion and exclusion criteria and will undergo the intervention.
  The subject will be randomly assigned to the three groups:
  a morning training group (n=14, 5 men, 9 women) an afternoon training group (n=14, 5 men, 9women) a control group (n=6, 6 women) Both men and women will be included to address the potential differences between sexes and to increase the clinical and practical relevance, since women make up more than 50 percent of clients visiting the Centre of Active Aging.
  The duration of the training intervention is 12 weeks with the frequency 2 times per week.
  The relative volume and intensity of the training for both training groups will be identical, except for timing of the training. The morning group and afternoon group will exercise exclusively between 08:00 - 09:00 h and 16:00 - 17:00 h, respectively.
Masking Description: Due to the time-specificity of the training design there is no possibility to mask the subject distribution.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Morning group (Experimental): The experimental factor will be applied in the morning (8:00-9:00).
  Interventions: Procedure: Combined training
- Afternoon group (Experimental): The experimental factor will be applied in the afternoon (16:00-17:00).
  Interventions: Procedure: Combined training
- Control group (No Intervention): None expertimental factor will be aplied

INTERVENTIONS:
Procedure: Combined training — 12-week long time specific combined training 2 times a week
  Arms: Afternoon group; Morning group

SUMMARY:
The project aims to explore the mechanisms, by which physical activity can support healthy ageing and decrease the negative impact of ageing on the circadian system, musculoskeletal system and immunity.

DETAILED DESCRIPTION:
The main aim of the project is to examine the effect of as well as of the three-month, timely specific training intervention on the functionality of circadian organization in elderly volunteers. The additive aim is to examine the effect of lifelong endurance physical activity, along with the experimental training intervention on the body composition, bone density, and selected hormonal, biochemical, histological and molecular indicators of metabolic health.

Partial aims are as follows:n to explore the effect of morning and afternoon training on the most significant parameters, identified by the previous cross-sectional study, in sedentary elderly. Furthermore, to clarify adaptation mechanisms of experimental training protocol on selected parameters, that may explain possible differences in mechanisms of active and passive aging.

ELIGIBILITY:
Inclusion Criteria:

* no history of regular physical activity training and exercise of more than 150 minutes of moderate or 75 minutes of higher intensity per week.
* Body mass index (BMI) between 18.5 and 30 kg/m2 for all groups

Exclusion criteria for probands will be:

* Recent or current infection, physical disability,
* malignant, cardiovascular, metabolic, autoimmune diseases,
* Malnutrition and pharmacological interference (e.g., steroids, non-steroidal anti-inflammatory agents, immunosuppressive and antineoplastic drugs).

Use of performance enhancing drugs in the past and during the study period will condition exclusion.

Exclusion Criteria:

* recent or current infection, physical disabilities,
* malignant, cardiovascular, metabolic, autoimmune diseases,
* Malnutrition and pharmacological interference (e.g., steroids, nonsteroidal anti-inflammatory agents, immunosuppressive and antineoplastic drugs).

Use of performance-enhancing drugs in the past and during the study period will condition exclusion.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 34 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-07-04 (Actual); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Bone mineral density | 12 weeks
  The proportion of total body fat mass, visceral fat mass, total body mass and bone density will be measured using Dual-energy X-ray Absorptiometry (DXA, hologic fan-beam bone densitometer Discovery QDR series). The DXA testing procedure will follow Kralik et al. (2019). All DXA procedures will be performed by a board-certified radiologist.

CONTACTS AND LOCATIONS:
Locations (1):
- Comenius University in Bratislava, Faculty of physical education and sport Bratislava, Slovakia, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-16): https://cdn.clinicaltrials.gov/large-docs/49/NCT06746649/Prot_SAP_000.pdf